CLINICAL TRIAL: NCT02204267
Title: Impact of Standardized MONitoring for Detection of Atrial Fibrillation in Ischemic Stroke
Acronym: MonDAFIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Principal Investigator, Matthias Endres, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MonDAFIS; EA2/033/14 (Other: Ethics comission, Charité)
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Stroke; atrial fibrillation; ECG
MeSH Terms: conditions — Stroke; Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prolonged ECG monitoring (Experimental): Regular stroke unit treatment and diagnostic procedures according to guidelines and additional prolonged ECG monitoring
  Interventions: Other: prolonged ECG monitoring; Device: ECG
- no additional ECG recording (No Intervention): Regular stroke unit treatment and diagnostic procedures according to guidelines

INTERVENTIONS:
Other: prolonged ECG monitoring — Start of long-term ECG immediately after admission to the stroke unit by using a portable ECG recorder for a max. duration of 7 days (or hospital discharge)
  Arms: prolonged ECG monitoring
Device: ECG
  Arms: prolonged ECG monitoring

SUMMARY:
Investigator-initiated prospective randomized multicentre study to uncover the true burden of paroxysmal atrial fibrillation in a representative population of acute stroke patients without known atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke or transitory ischemic attack (with clinical deficit on enrolment or MRI detected acute brain lesion on admission)
* Age ≥ 18 years
* Written or oral informed consent
* Stroke unit admission within 72 hours after stroke onset
* Start of standardized prolonged ECG monitoring within 24 hours after admission to the stroke unit
* Willingness to take part in the planned follow up examinations

Exclusion Criteria:

* Known atrial fibrillation
* Atrial fibrillation detected by ECG on admission
* Atrial fibrillation detected prior study enrollment on the stroke unit
* Life expectancy < 1 year (before actual stroke)
* Life expectancy < 1 month (after actual stroke)
* Indication for oral anticoagulation other than atrial fibrillation (e.g. mechanical heart valve)
* Severity level according National Institute of Health Stroke Scale (NIHSS) score > 22
* Participation in an interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3470 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Number of patients on oral anticoagulation (NOAC or VKA) | 12 months
  Number of study patients on oral anticoagulation (NOAC or VKA) at 12 months after the index stroke either randomized to standardized prolonged ECG monitoring in-hospital or those randomized to usual stroke unit diagnostic procedures alone.

SECONDARY OUTCOMES:
Number of stroke patients with newly detected atrial fibrillation | 7 days
  Number of stroke patients with newly detected atrial fibrillation using a standardized prolonged ECG monitoring compared to usual stroke unit diagnostic procedures alone.

OTHER OUTCOMES:
Impact of stroke unit level on the rate of atrial fibrillation detection | 7 days
  Impact of stroke unit level (i.e. primary or comprehensive stroke center) on the rate of atrial fibrillation detection in-hospital stroke in patients randomized to standardized prolonged ECG monitoring in hospital
Number of recurrent strokes, major bleeds, myocardial infarction and all-cause death (composite endpoint) within 6, 12 and 24 months after the index stroke | 24 months
  Number of recurrent strokes, major bleeds, myocardial infarction and all-cause death (composite endpoint) within 6, 12 and 24 months after the index stroke in patients either randomized to standardized prolonged ECG monitoring in-hospital or those randomized to usual stroke unit diagnostic procedures alone.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Endres, MD, Principal Investigator — Center for Stroke Research Berlin, Charité University Berlin, Campus Mitte
Locations (1):
- Charité Universitaetsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Haeusler KG, Tutuncu S, Fiessler C, Jawad-Ul-Qamar M, Kunze C, Schurig J, Dietzel J, Kramer M, Petzold GC, Royl G, Helberg T, Thomalla G, Nabavi DG, Rother J, Laufs U, Veltkamp R, Heuschmann PU, Kirchhof P, Olma MC, Endres M. Excessive Supraventricular Ectopic Activity in Patients With Acute Ischemic Stroke Is Associated With Atrial Fibrillation Detection Within 24 Months After Stroke: A Predefined Analysis of the MonDAFIS Study. J Am Heart Assoc. 2025 Jan 21;14(2):e034512. doi: 10.1161/JAHA.123.034512. Epub 2025 Jan 10. PMID 39791425
- [Derived] Tutuncu S, Olma MC, Kunze C, Dietzel J, Schurig J, Rosenkranz M, Stingele R, Maschke M, Heuschmann PU, Kirchhof P, Laufs U, Nabavi DG, Rother J, Thomalla G, Veltkamp R, Endres M, Haeusler KG; MonDAFIS Investigators. Heart failure, recurrent vascular events and death in patients with ischemic stroke-results of the MonDAFIS study. Intern Emerg Med. 2024 Aug;19(5):1247-1254. doi: 10.1007/s11739-024-03594-8. Epub 2024 Apr 15. PMID 38619714
- [Derived] Ingwersen T, Olma MC, Schlemm E, Mayer C, Cheng B, Tutuncu S, Kirchhof P, Veltkamp R, Rother J, Laufs U, Nabavi DG, Ntaios G, Endres M, Haeusler KG, Thomalla G. Independent external validation of a stroke recurrence score in patients with embolic stroke of undetermined source. Neurol Res Pract. 2023 Oct 5;5(1):51. doi: 10.1186/s42466-023-00279-z. PMID 37794453
- [Derived] Olma MC, Tutuncu S, Grittner U, Kunze C, Jawad-Ul-Qamar M, Kirchhof P, Rother J, Thomalla G, Veltkamp R, Laufs U, Nabavi DG, Heuschmann PU, Endres M, Haeusler KG. Extent of routine diagnostic cardiac work-up at certified German stroke units participating in the prospective MonDAFIS study. Neurol Res Pract. 2023 Jun 1;5(1):21. doi: 10.1186/s42466-023-00246-8. PMID 37259147
- [Derived] Olma MC, Tutuncu S, Fiessler C, Kunze C, Kramer M, Steindorf-Sabath L, Jawad-Ul-Qamar M, Kirchhof P, Laufs U, Schurig J, Kraft P, Rother J, Gunther A, Thomalla G, Dimitrijeski B, Nabavi DG, Veltkamp R, Heuschmann PU, Haeusler KG, Endres M; MonDAFIS Investigators [Link]. In-Hospital ECG Findings, Changes in Medical Management, and Cardiovascular Outcomes in Patients With Acute Stroke or Transient Ischemic Attack. J Am Heart Assoc. 2023 Jan 17;12(2):e027149. doi: 10.1161/JAHA.122.027149. Epub 2023 Jan 11. PMID 36628982
- [Derived] Haeusler KG, Kirchhof P, Kunze C, Tutuncu S, Fiessler C, Malsch C, Olma MC, Jawad-Ul-Qamar M, Kramer M, Wachter R, Michalski D, Kraft A, Rizos T, Groschel K, Thomalla G, Nabavi DG, Rother J, Laufs U, Veltkamp R, Heuschmann PU, Endres M; MonDAFIS Investigators. Systematic monitoring for detection of atrial fibrillation in patients with acute ischaemic stroke (MonDAFIS): a randomised, open-label, multicentre study. Lancet Neurol. 2021 Jun;20(6):426-436. doi: 10.1016/S1474-4422(21)00067-3. PMID 34022169
- [Derived] Haeusler KG, Kirchhof P, Heuschmann PU, Laufs U, Busse O, Kunze C, Thomalla G, Nabavi DG, Rother J, Veltkamp R, Endres M. Impact of standardized MONitoring for Detection of Atrial Fibrillation in Ischemic Stroke (MonDAFIS): Rationale and design of a prospective randomized multicenter study. Am Heart J. 2016 Feb;172:19-25. doi: 10.1016/j.ahj.2015.10.010. Epub 2015 Oct 21. PMID 26856211